CLINICAL TRIAL: NCT03941561
Title: Compare S-1 for 9 Months to 1 Year as Adjuvant Chemotherapy in Stage II Gastric Cancer (SMAC）
Brief Title: S-1 for 9 Months Versus 1 Year for Stage II Gastric Cancer (SMAC）
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGCG006
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; S-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Tegafur; gimeracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-1 for 9 months (Experimental): S-1 80-120mg daily for 14 days in 3 weeks for totally 9 months after D2 resection
  Interventions: Drug: S-1 for 9 months
- S-1 for 1 year (Active Comparator): S-1 80-120mg daily for 14 days in 3 weeks for totally 1 year after D2 resection
  Interventions: Drug: S-1 for 1 year

INTERVENTIONS:
Drug: S-1 for 9 months — S-1 for 9 months after D2 resection
  Other Names: Tegafur,Gimeracil and Oteracil Porassium Capsules
  Arms: S-1 for 9 months
Drug: S-1 for 1 year — S-1 for 1 year after D2 resection
  Other Names: Tegafur,Gimeracil and Oteracil Porassium Capsules
  Arms: S-1 for 1 year

SUMMARY:
The study aims to compare the efficacy and safety of S-1 for 9 months versus S-1 for 1 year as adjuvant chemotherapy after D2 resection in patients with gastric cancer.

Hypothesis: For gastric patients after D2 resection, S-1 for 9 months shows non-inferiority to S-1 for 1 year in disease-free survival(DFS), overall survival (OS) and safety.

DETAILED DESCRIPTION:
It has been identified that S-1 is an effective adjuvant treatment for East Asian patients who have undergone a D2 dissection for locally advanced gastric cancer（GC) in the Japanese Adjuvant Chemotherapy Trial of TS-1（S-1) for Gastric Cancer (ACTS-GC) trail, And S-1 has become one of the standard therapies to these patients. But it is still unknown whether it would improve equally or even more to overall survival(OS) and disease-free survival(DFS) than S-1 for 1 year compared with S-1 for 9 months. As a result, An further clinical trial is still needed, This trial is designed to investigate the efficacy and safety of S-1 for 9 months versus S-1 for 1 year as adjuvant chemotherapy after D2 resection in patients with gastric cancer.

In this study, patients histologically confirmed stage II and who received D2 resection were randomly assigned to receive S-1 for 9 months or S-1 for 1 year. Patients aged from 18 to 75 years and adequate organ function are randomized 1:1 to S-1 for 9 months and S-1 for 1 year. Both are the 3-week recycle of S-1 (80-120mg per day) for 2 weeks, followed by 1 week of rest. The primary endpoint is 3-year DFS, and the secondary endpoint is 5-year OS and safety. Final study analysis will be conducted at the end of the 5th year after the last patient's enrollment. In summary, we hold the hypothesis that S-1 for 9 months is equally effective, safer, and easier to carry out. If possible, there will be a new adjuvant chemotherapy strategy for gastric cancer patients after D2 resection.

To ensure the quality of the study, two interim analyses will be planned at the half and the completion of the study respectively. The DATA and Safety Monitoring Committee will independently review the interim analysis and stop the study ahead of schedule if necessary. Furthermore, to improve the study progress and quality, the in-house interim monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. The lower age limit of research subjects 18 years old and upper age limit of 75 years old.
2. Be proven to be primary adenocarcinoma of gastric cancer and staged II by pathological evidence
3. R0 surgery with lymphadenectomy
4. Without any other malignancies
5. ECOG (ECOG score standard) performance status of 0 or 1 and expected to survive more than 6 months
6. No contraindications to chemotherapy, including normal peripheral blood routine, liver, and kidney function and electrocardiogram （WBC≥4.0 x 109 /L, NEU≥1.5 x 109 /L, PLT≥100 x 109 /L and HGB≥90g/L).

Exclusion Criteria:

1. Female in pregnancy or lactation, or refuse to receive Contraception measures during chemotherapy.
2. Patients with stage I, III and IV.
3. Unavailable for R0 resection and D2 lymph node dissection.
4. Suffering from other uncontrolled diseases, such as other tumors, acute and Chronic infection.
5. With severe heart disease, including congestive heart failure, uncontrolled arrhythmias, unstable angina, myocardial infarction, severe heart valve disease, and resistant hypertension.
6. Any Known or suspected history of drug allergy test.
7. The researchers believe the patient is not able to complete the entire course of the experiment.
8. Patients (within 4 weeks) are receiving any other anti-cancer drugs therapy, biological therapy, radiation therapy, or Immunosuppressive therapy.
9. Patients conform to any of the following: post-organ transplant, necessary for long-term immunosuppressive or suffering with autoimmune diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
DFS | 3-year
  Disease-free survival

SECONDARY OUTCOMES:
OS | 5-year
  Overall survival

OTHER OUTCOMES:
Side effects | 1-year
  Complications such as Nausea, vomiting, myelosuppression, and Liver or kidney function disorder

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, PHD, MD, Principal Investigator — Fudan University
Locations (6):
- China (6):
  - Anqing Municipal Hospital, Anqing
  - Second Affiliated Hospital, School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Jiangxi Provincial Cancer Hospital, Nanchang
  - Dazhi Xu, Shanghai
  - First Affiliated Hospital of Wannan Medical College, Wuhu